CLINICAL TRIAL: NCT06145464
Title: Shadow for All, a Citizenship Science Study to Promote the Prevention of Skin Cancer
Acronym: Shadow4All
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Shadow4All
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-11

CONDITIONS: Skin Cancer
Keywords: skin cancer; prevention; adolescents; literacy; citizen science
MeSH Terms: conditions — Skin Neoplasms; Literacy

STUDY DESIGN:
Intervention Model Description: Exploratory pilot study, with a quasi-experimental design
Who Masked: Participant
Masking Description: The target population will be single-blinded towards the professional activity of providers of health literacy sessions about the prevention of skin cancer in the two interventional groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Adolescents will be recommended to use the sun protection interventions implemented on Foz do Lizandro beach (collective shadow, sun protector, and information about healthy behaviors of sun protection disposed in an infographic installed near the collective shadow), without a previous health literacy session about skin cancer prevention provided 15 days before the beginning of the use of the interventions on the beach.
  Interventions: Behavioral: Adhesion to the use of collective shadow; Behavioral: Adhesion to the use of sun protector; Behavioral: Adhesion to the use of the information disposed in the infographic
- Interventional EST SUP (Experimental): Adolescents will be recommended to use the sun protection interventions implemented on Foz do Lizandro beach (collective shadow, sun protector, and information about healthy behaviors of sun protection disposed in an infographic installed near the collective shadow), with a previous health literacy session about skin cancer prevention provided 15 days before the beginning of the use of the interventions on the beach by students on ongoing graduation at the University of Lisbon.
  Interventions: Behavioral: Adhesion to the use of collective shadow; Behavioral: Adhesion to the use of sun protector; Behavioral: Adhesion to the use of the information disposed in the infographic; Behavioral: Adhesion to the health literacy sessions in the interventional groups
- Interventional FARMA (Experimental): Adolescents will be recommended to use the sun protection interventions implemented on Foz do Lizandro beach (collective shadow, sun protector, and information about healthy behaviors of sun protection disposed in an infographic installed near the collective shadow), with a previous health literacy session about skin cancer prevention provided 15 days before the beginning of the use of the interventions on the beach by community pharmacists who will be working on pharmacies located in Mafra.
  Interventions: Behavioral: Adhesion to the use of collective shadow; Behavioral: Adhesion to the use of sun protector; Behavioral: Adhesion to the use of the information disposed in the infographic; Behavioral: Adhesion to the health literacy sessions in the interventional groups

INTERVENTIONS:
Behavioral: Adhesion to the use of collective shadow — Quantitative evaluation of the use of shadow provided by one or two collective fabric devices, with 6 per 3 metres of size, containing 100% UV blocking filters, that will be installed in the sand on Foz do Lizandro beach, according to the recommendations provided in all groups of the study.
Behavioral: Adhesion to the use of sun protector — Quantitative evaluation of the use of sun protector according to the recommendations provided in all groups of the study.
Behavioral: Adhesion to the use of the information disposed in the infographic — Quantitative evaluation of the use of the information disposed in the infographic and provided in all groups of the study.
Behavioral: Adhesion to the health literacy sessions in the interventional groups — Provision of health literacy sessions about skin cancer prevention by two different types of providers in the two interventional groups, 15 days before the use of sun protective interventions implemented at the beach
  Arms: Interventional EST SUP; Interventional FARMA

SUMMARY:
The proposed project is a pilot study about the impact of different health literacy interventions, focused on preventing skin cancer, on the adhesion to protection strategies against ultraviolet (UV) radiation, observed in high school students, that will be implemented on Foz do Lizandro beach in the municipality of Mafra, Portugal. As a science project with citizenship and respecting the ethic principles of equity, inclusion and diversity, the study will involve the contribution and participation of institutional and community partners in diverse stages of the research study: design, field implementation, data collection and dissemination of results, as well as financial investment for the acquisition and installation of interventions on the beach, and recruitment of the target population.

DETAILED DESCRIPTION:
The incidence of skin cancer has increased very fast globally, largely due to poor protective behavior against highly harmful UV solar radiation, particularly among the Caucasian population, who are the most affected by this type of cancer. Scientific literature suggests that adolescents between14 and 17 years old are very susceptible to getting sunburned at least once, which doubles the risk of developing skin cancer in adulthood. It is also known that literacy about skin cancer and its prevention is not high in these younger age groups. These data suggest that the design of public health policies aimed at adolescents, focused on promoting healthy habits of exposure to solar and artificial UV radiation, should be a priority.

Based on this scientific evidence, a quasi-experimental and interventional pilot study is proposed, through which the aim is to motivate adolescents between 14 and 17 years old to adhere to the use of sun protection strategies to be implemented on Foz do Lizandro beach in municipality of Mafra, Portugal.The research question is to understand whether different literacy sessions on skin cancer prevention have a different impact on adhesion to sun protection strategies used by participating adolescents. Considering the enormous potential of the study to become a science project with citizenship, its design was adapted to this increasingly valued modality of research, so that local community entities and national institutions are part of the study as individual and collective partners, participating in the various stages of the investigation, from structuring, implementation in the field, analysis and dissemination of results. Values such as equity, inclusion, diversity and sustainability are inherent to the study. Monitoring of project implementation will be done through the determination of rigorously planned quality indicators.

It is expected that this study will have a positive impact on Mafra community and will be replicated in other geographic regions, leading to significantly higher literacy levels on skin cancer prevention among the youngest citizens.

ELIGIBILITY:
Inclusion Criteria for adolescents

* High school students at a public school in Mafra;
* Age between 14 and 17 years old;
* Residents in Mafra;
* Fluent in the Portuguese language;
* Regular users of beaches in the summer season

Exclusion Criteria for adolescents

* Cognitive, hearing, visual and/or motor limitations that prevent the acquisition of knowledge and the use of sun protection strategies on the beach

Inclusion Criteria for universitarian students

* Students at a higher education course in the area of health sciences;
* Age between 18 and 25 years old;
* Motivated to the field of health communication;
* Preferably, with experience in research work during the course.

Exclusion Criteria for universitarian students

* Cognitive, hearing, visual and/or motor limitations that prevent the acquisition and transmission of knowledge

Inclusion Criteria for community pharmacists

* Professionally active in a community pharmacy in the region where the beach is located;
* Preferably young people between 23 and 45 years old, regardless of professional experience;
* With motivation for awareness-raising activities on disease prevention in communities;
* Preferably, who have already carried out this type of awareness-raising actions among younger people on disease prevention or, specifically, on the prevention of skin cancer;
* Affinity for the topic of skin cancer and its prevention.

Exclusion Criteria for community pharmacists

* Cognitive, hearing, visual and/or motor limitations that prevent the acquisition and transmission of knowledge

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Adhesion to the use of sunsail shadows | 2 months (July + August 2024)
  Number of adolescents who use the sunsail shadows among all participant adolescents, in all groups of the study
Adhesion to the use of sunscreen | 2 months (July + August 2024)
  Number of adolescents who adhere to the use of sunscreen among all participant adolescents, in all groups of the study
Adhesion to the use of infographic´s information | 2 months (July + August 2024)
  Number of adolescents who read and use the information related to the promotion of healthy sun exposure behaviors, from the infographic located near the sunsail shadows, in all groups of the study
Adhesion to the use of interventional strategies of sun protection at the beach | 2 months (July + August 2024)
  Number of adolescents who use one, two or all of the three interventional strategies of sun protection implemented at the beach, in all groups of the study
Skin absorption of UV radiation | 2 months (July + August 2024)
  Number of adolescents who have a safe skin UV radiation absorption according to the interventional sun protection strategies used, in all groups of the study
Impact of literacy sessions about the prevention of skin cancer on the amount of skin UV absorption in all interventional groups compared to the control group | 2 months (July + August 2024)
  Amount of skin UV absorption per total number of participant adolescents in both interventional groups, in relation to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Magda Fonseca, Master, Principal Investigator — RD-Portugal (Rare Diseases-Portugal)

IPD SHARING:
Plan to Share IPD: No